CLINICAL TRIAL: NCT02314286
Title: Rosuvastatin Use in Order to Induce Preeclampsia Resolution in Severe Preeclampsia Cases up to 48 Hours Following Delivery
Brief Title: Rosuvastatin in Order to Induce Preeclampsia Resolution in Severe PET up to 48 Hours Following Delivery
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Ofer Beharier, Physician at Obstetrics and Gynecology Division, Soroka University Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: sor005514ctil; SCRC14001 (Other: soroka)
Record Dates: First submitted 2014-11-16; First posted 2014-12-11 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Severe Pre-eclampsia
Keywords: Rosuvastatin; severe preeclampsia; 48 hours following delivery
MeSH Terms: conditions — Pre-Eclampsia | interventions — Rosuvastatin Calcium; AtpH protein, E coli

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (Placebo Comparator): After signing an informed consent form and filling a demographic and medical questionnaire, a randomization 1:1 will be carried. 50 women will be in the control arm. the group will be treated according to ACOG guidelines (Appendix). After the delivery, a small placenta sample will be collected.
  Control group will be treated with placebo.
  Interventions: Drug: Placebo
- treatment (Experimental): 50 women will be in the treatment arm. the group will be treated according to ACOG guidelines (Appendix). After the delivery, a small placenta sample will be collected. In addition, following randomization experimental group will be treated with Rosuvastatin 40mg that will be administrated orally with or without food. Treatment will be carried within the first hour following delivery. Another dose will be given 24 hours after first administration. Control group will be treated with placebo.
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin is a hydrophilic statin, short treatment (hours to days) with this type of statin improved the outcome of patients during acute myocardial infarction, sepsis, contrast-induced nephropathy, hepatic ischemia/reperfusion injury, emphasizing its preferential pleiotropic effects. Currently, the FDA classiﬁes all statins as pregnancy category X and discourages their use during pregnancy due to higher abortion rate and teratogenicity that were observed in animals exposed to hydrophobic statins during pregnancy. Since the use of statins after delivery is allowed, the present study will aim to evaluate whether Rosuvastatin may accelerates preeclampsia resolution following delivery and potentially reduce postpartum preeclampsia complications.
  Other Names: Stator
  Arms: treatment
Drug: Placebo
  Arms: control

SUMMARY:
Prospective randomized single blind trial. Study population are women diagnosed with severe pre-eclampsia during singleton pregnancy, between 24+0 weeks and 41+6 weeks gestational age. The purpose of the study is to evaluate the effect of Rosuvastatin on the severe preeclampsia resolution at 48 hours after delivery. After screening and signing an informed consent form, before entering delivery room, a randomization 1:1 will be carried. 50 women will be in the treatment arm while 50 will be in the control arm. Both groups will be treated according to ACOG (The American College of Obstetricians and Gynecologists has the following clinical guidelines related to deliveries before 39 weeks) guidelines. In addition, following randomization experimental group will be treated with Rosuvastatin 40mg that will be administrated orally with or without food. Treatment will be carried within the first hour following delivery. Another dose will be given 24 hours after first administration. Control group will be treated with placebo.

DETAILED DESCRIPTION:
Preeclampsia is a disorder of widespread vascular endothelial malfunction and vasospasm that occurs after 20 weeks' gestation and can present as late as 4-6 weeks' postpartum. It is clinically defined by as blood pressure ≥140 mmHg systolic and ≥90 mmHg diastolic diagnosed for the first time after 20 weeks' gestation together with >300mg proteinuria/24 hours.

The global incidence of preeclampsia has been estimated at 5-14% of all pregnancies. Pre-eclampsia affects approximately 6-8% of all pregnancies worldwide. Pre-eclampsia affects 3-5% of all first time pregnancies, but early severe pre-eclampsia occurs in only 1:200 pregnancies.

Significant risk factors for pre-eclampsia are as follows: Nulliparity, age >40 years, black race, family history, chronic renal disease, chronic hypertension, antiphospholipid syndrome, diabetes mellitus , multiple gestation and high body mass index.

Mild preeclampsia is defined as the presence of hypertension (BP ≥140/90 mm Hg) on 2 occasions, at least 6 hours apart, but without evidence of end-organ damage.

Severe preeclampsia is defined as the presence of 1 of the following symptoms or signs in the presence of preeclampsia:

marked elevation of blood pressure (>160/110 mmHg), severe proteinuria (>5 g/24 hours), or evidence of central nervous system (CNS) dysfunction (headaches, blurred vision, seizures, coma), renal dysfunction (oliguria or creatinine > 1.5 mg/dL), pulmonary edema, hepatocellular injury (ALT > 2-fold the upper limits of normal), hematologic dysfunction (platelet count < 100,000/L or DIC), or placental dysfunction (oligohydramnios or severe intrauterine growth restriction). The HELLP (hemolysis, elevated liver enzymes, low platelets) syndrome is a special subgroup of severe preeclampsia and is a major cause of morbidity and mortality.

Eclampsia is defined as seizures that cannot be attributable to other causes in a woman with preeclampsia.

The optimal management of a woman with preeclampsia depends on gestational age and disease severity Management of preeclampsia is challenging because it requires the clinician to balance the health of the mother and fetus simultaneously. Patients with mild preeclampsia are often induced after 37 weeks gestation. Before this, the immature fetus is treated with expectant management with bed rest, close monitoring of blood pressure and renal function, and careful fetal surveillance. For women with severe preeclampsia, induction of delivery should be considered after 34 weeks gestation unless the patient is eligible for expectant management in a tertiary hospital setting. The definitive treatment of preeclampsia is delivery of the fetus and placenta. Anti-hypertensive drugs are essential for severe hypertension (≥160 mmHg systolic or ≥110 mmHg diastolic) for reducing the risk of cerebrovascular accidents. Intravenous Labetalol, Nifedipine or hydralazine are the drugs most commonly used to manage preeclampsia but there is insignificant evidence to indicate which drug is preferable..

Magnesium sulfate is the treatment of choice for the prevention and treatment of eclamptic seizures Where immediate child-birth is not essential, a delay of 24 hours will allow steroids to be given to mature the baby's lungs, although a shorter duration may still be of benefit.

Preeclampsia is associated with short-term and long-term maternal and fetal complications. For the mother, it may lead to eclamptic seizures, stroke, intracranial bleed, uncontrolled hypertension, renal failure, and hemolysis. For the fetus, it may lead to intrauterine growth restriction, placental abruption, and the short-term and long-term complications of prematurity, as well as predisposition to adult cardiovascular and metabolic disorders. Currently, there is no effective therapy to preeclampsia, and delivery remains the only approach to preventing maternal morbidity and mortality. However, this is usually achieved at the expense of premature delivery and its associated morbidities. Moreover, following the delivery, preeclampsia resolved slowly within days, exposing the mother to late complications and increasing treatment cost significantly.

To date, the exact etiology of preeclampsia remains unknown. However, evidence obtained in recent years, supports the theory that angiogenic imbalance is the end common pathway that leads to clinical preeclampsia. During normal pregnancy, vascular endothelial growth factor (VEGF) and placental growth factor (PlGF) promote pro-angiogenic state that regulates vascular tone and glomerular capillary health. In preeclampsia, these proteins are antagonized by excessive placental production of soluble fms-like tyrosine kinase-1 (sFlt-1), thereby creating angiogenic imbalance. After delivery, this imbalance resolves within hours to days correlating with the resolution of the disease. One of the observations that marked sFlt-1 as key player in the pathogenesis of preeclampsia was made in an animal model. It was demonstrated that preeclampsia can be induced in animal model by over expressing sFlt-1 alone. In their model hydrophilic statins treatment decreased sFlt-1 levels and up-regulated VEGF and PlGF levels. Most importantly, statins ameliorated preeclampsia symptoms by improving hypertension and proteinuria in the preeclamptic mice.

Statins are potent inhibitors of cholesterol biosynthesis and used successfully in the primary and secondary prevention of coronary heart disease. Additionally, statins are known to mediate pleiotropic effects via improving endothelial function and attenuating inflammatory responses. Rosuvastatin is a hydrophilic statin, characterized by low permeability through membranes, as the placenta and blood-brain-barrier. In addition, Short treatment (hours to days) with this type of statin improved the outcome of patients during acute myocardial infarction, sepsis, contrast-induced nephropathy, hepatic ischemia/reperfusion injury, emphasizing its preferential pleiotropic effects.

Currently, the food and drug administration classiﬁes all statins as pregnancy category X and discourages their use during pregnancy due to higher abortion rate and teratogenicity that were observed in animals exposed to hydrophobic statins during pregnancy. Evidence for teratogenicity of the hydrophilic statins was never reported probably due to their limited permeability across membranes. Since the use of statins after delivery is allowed, the present study will aim to evaluate whether Rosuvastatin may accelerates preeclampsia resolution following delivery and potentially reduce postpartum preeclampsia complications.

ELIGIBILITY:
Inclusion Criteria:

1. Women who understand and sign the informed consent form.
2. Women over the age of 18.
3. Women between 24+0 weeks and 41+6 weeks gestation
4. Women with singleton viable pregnancy.
5. Have a diagnosis of severe pre-eclampsia

Exclusion Criteria:

1. Eclampsia (convulsions)
2. Current use of statins
3. Women during active labor (5 cm and above)
4. Contraindications to statin use (other than pregnancy) including:

   * Hypersensitivity to Rosuvastatin or any of its excipients
   * Active liver disease or elevation of serum Transaminases >3 ULN) believed to be unrelated to pre- eclampsia.
   * Pre-pregnant renal insufficiency (creatine clearance less than 30 ml/min)
   * Concomitant administration of medications known to interact with Rosuvastatin (e.g. Cimetidine)
5. A known or suspected adverse reaction in former statin use.
6. Transfer to a non-trial centre
7. Women who would like to breastfeed 24-48 hours after delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of Rosuvastatin on the severe preeclampsia resolution at 48 hours after delivery | 48 hours

SECONDARY OUTCOMES:
Time from delivery until reduction in general blood pressure | 48 hours
  systolic pressure below 140mm\Hg or diastolic pressure below 90mm\Hg. Measurement will be carried out according to standard Protocol: before delivery, every 30 minutes during the first 2 hours post-delivery then every hour until discharge.
Duration and dosage of hypertensive treatment due to severe hypertension (systolic greater than 160 mmHg or diastolic greater than 110 mmHg | 48 hours
Evaluation of renal function through urine Protein / creatinine ratio measurement will be examined before delivery and 6, 12, 18, 24 hours post-delivery. In addition the time from delivery to polyuria will be assessed via measuring urine output per hour. | 48 hours
Rate of liver transminases resolution. Samples will be taken before delivery and every 6 hours post-delivery (part of the routine follow-up of preeclampsia). | 48 hours
Examining time to thrombocytopenia resolution. Samples will be taken before delivery and every 6 hours post-delivery (part of the routine follow-up of preeclampsia). | 48 hours
Length assessment of intensive care unit hospitalization | 48 hours and beyond
Immunological assessment of the placenta | 48 hours and beyond
  We intend to test the following metrics:
  1. The amount and activity of NK cells in the placenta.
  2. The rate of secretion of angiogenic factors VEGF, SFLT-1, PLGF and inflammation factors TGF-ALFA I and IL-6.